CLINICAL TRIAL: NCT00535379
Title: SUTENT (SUNITINIB, SU11248)in Patients With Recurrent or Progressive Glioblastoma Multiforme An Academic Prospective Single-arm Phase II Clinical Trial Including Ranslational Research Studies
Brief Title: SUTENT (SUNITINIB, SU11248)in Patients With Recurrent or Progressive Glioblastoma Multiforme
Acronym: SURGE01-07
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Medical University Innsbruck, Department of Neurology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT-Nr. 2007-002142-37
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2009-01

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme; sunitinib; recurrent; progressive
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients will receive SUTENT 37.5mg (3 x 12.5mg capsules) PO daily in the morning after breakfast. After 2 weeks without treatment-related adverse events grade ≥ 2 (ECOG common toxicity criteria: refer to Protocol Attachment A.4) a SUTENT dose escalation to 50mg (4 x 12.5mg capsules) PO daily has to be performed. Treatment will continue until patients develop progression of disease or until unacceptable adverse events occur.
  Other Names: SUTENT

SUMMARY:
Clinical Part:

The objective of this study is to determine the efficacy and safety of SUTENT in patients with recurrent or progressive glioblastoma multiforme.Patients with tissue based diagnosis of intracranial glioblastoma multiforme, above 18 years of age and of both genders, who have a first tumor recurrence or progress after surgery, radiation- and chemotherapy will be included. The hypothesis is that SUTENT will significantly increase the progression free survival rate at 6 months in the study population.

DETAILED DESCRIPTION:
Background Glioblastoma multiforme (GBM) is the most common and most aggressive primary brain tumor in adults and shows an incidence of 5/100.000 inhabitants per year1. In Austria, approximately 350 patients are diagnosed with malignant glioma annually. Advances in surgery, radiotherapy and chemotherapy do only have a minor impact on the natural course of these hardly treatable tumors. The mean survival time of adult patients with GBM is only 9-15 months from the time of diagnosis1,2. Thus, there is an urgent need for more effective therapeutic approaches based on a better molecular understanding of tumor progression and tumor neovascularization.

Molecular Neurooncology has begun to elucidate the complexity of the transformed phenotype of GBM with the goal to identify important molecular changes in the tumor cell that may be amenable for targeted therapies3.

The elucidation of growth factor receptor signaling pathways responsible for the malignant phenotype is now being translated into molecular therapies. At present, targeted therapies with small molecule inhibitors directed against receptor tyrosine kinases (RTKs) or downstream signaling pathways seem to be the most promising therapeutic approaches by directly influencing oncogenetically altered signaling pathways4. Imatinib Mesylate (STI571, Gleevec) is a potent inhibitor of the Bcr-Abl, PDGFR-α/ß, c-Fms and c-KIT tyrosine kinases. Its ability to inhibit PDGFR signaling suggested therapeutic potential in malignant gliomas, but single-agent imatinib showed only minimal therapeutic activity5. Erlotinib (OSI-774, Tarceva) and Gefitinib (ZD1839, Iressa) are potent inhibitors of the Epidermal-Growth-Factor-Receptor (EGFR). However, both inhibitors have also demonstrated only limited activity in GBMs with response rates of 10 to 15% and no significant prolongation of survival6. Tipifarnib (R115777, Zarnestra) is a potent and selective inhibitor of the farnesyl-transferase and influences the Ras oncogene pathway. Overexpression of Ras is implicated in the pathogenesis of malignant gliomas, but also amplified receptors as EGFR, PDGFR and VEGFR can lead to its downstream activation. Clinical trials with inhibition of the Ras signaling pathway showed also only limited biologic effects in GBM patients7.

3.2. Rationale for SUTENT treatment of GBM Patients Reason for the limited activity of selective targeting single agents, but also chemotherapeutic treatments, in GBM patients is the heterogeneity and redundancy of the molecular pathways in glioma cells8. Therefore, a multi-targeted therapy approach, inhibiting multiple molecular signaling pathways involved in tumor progression and tumor neovascularization seems to be a more promising treatment strategy.

SUTENT (SUNITINIB, SU11248) is a potent multi-target inhibitor of VEGFR1-3, PDGFR-α/β, FLT3, c-KIT, RET and CSF-1R. This drug has shown good solubility, bioavailability and protein-binding characteristics9 and was highly effective in metastatic clear-cell renal cell carcinoma (MRCC)10-12 and gastrointestinal stromal tumor (GIST)13,14.

The aggressiveness of GBM is reflected by a diffuse local infiltration into the brain parenchyma and a high tumor vascularization15,16. Neuropathological hallmarks of GBMs are pseudopalisades and microvascular hyperplasia. Pseudopalisades are characterized by an accumulation of hypoxic tumor cells around a central necrosis (Fig. 3A), resulting from increased metabolic demands of tumor cells or vascular occlusion. Such tumor cells express high levels of hypoxia-inducible regulators of angiogenesis, including the hypoxia-inducible factor (HIF)-α. HIF-α accumulates in the tumor cell and binds with its constitutively present partner HIF-β. The HIF complex leads to transcription of hypoxia-induced genes, such as VEGF and PDGF17. These growth factors are secreted into the extracellular space by tumor cells and bind to its high-affinity receptors located on

1. tumor cells (autocrine action), leading to tumor cell proliferation and survival, but also stimulation of the HIF-α protein synthesis and
2. endothelial cells, vascular smooth muscle cells and pericytes (paracrine action), leading to tumor-related neoangiogenesis18-21.

Therefore, VEGF may induce microvascular hyperplasia (Fig. 1B), a typical form of neoangiogenesis immediately related to pseudopalisading cells16,22. Since necrosis and hypoxia are located in the GBM's core, the most biologically relevant hypoxia-induced neovascularization occurs further peripherally, favouring diffuse infiltration by individual glioma cells and allows peripheral GBM expansion.

Summary of molecular and clinical rationales for SUTENT treatment of GBM patients

* The target molecules of SUTENT (i.e. VEGFR, PDGFR, FLT-3, c-KIT, RET) are strongly expressed in GBM tissue and have a crucial role in tumor progression and tumor neovascularization
* The vascular density in GBMs is among the highest of all human neoplasm
* Clinical studies with SUTENT demonstrated a radiological response and a significant improvement in progression free survival due to SUTENT treatment in MRCC and Imatinib-resistant GIST
* In clinical trials using SUTENT the incidence and severity of adverse events and laboratory abnormalities was relatively low (MRCC and GIST patients)

ELIGIBILITY:
Inclusion Criteria:

* Patients present with a first recurrence or first progression of a histological confirmed primary supratentorial glioblastoma multiforme WHO Grade IV (Classification following WHO criteria).
* Patients with surgical resection of first tumor progression: Following standard therapy patients must have evidence of first tumor progression. In general, patients may have undergone prior surgical resection of the first tumor progression and will be eligible if the following conditions apply:
* Patients must have recovered from the effects of surgery
* To adequately asses the GBM before surgery and the extent of residual disease postoperatively, two MRIs scans have to be performed:
* The first MRI scan within 2 weeks before surgery to document a progressed or recurrent GBM. The second MRI scan within 48 hours after surgery.
* Patients without surgical resection of first tumor progression:
* Patients must have evidence of first tumor progression following standard therapy as measured by a baseline MRI within 2 weeks prior to study enrollment (Macdonald criteria: i.e. tumor growth > 25% or new lesion).
* Resolution of all acute toxic effects of prior therapy to grade ≤ 1 (except alopecia)
* Patients must have an ECOG performance status of 0-2
* Patients must be ≥ 18 years and ≤ 75 years of age, with a life expectancy of greater than 8 weeks
* Patients must have adequate organ function as defined by the following criteria:

Bone Marrow Reserve - Platelets ≥ 75.000/μL

* Absolute Neutrophil Count (ANC) ≥ 1500/μL
* Hemoglobin ≥ 10.0 g/dL Blood Coagulation - aPTT ≤ 1.5 times upper limit of normal (ULN) Hepatic Function - ASAT and ALAT ≤ 1.5 times ULN
* ALP ≤ 2.5 times ULN
* Total Serum Bilirubin < 1 times ULN Renal Function - Serum Creatinine ≤ 1.5 times ULN Metabolism - Serum Albumin ≥ 3.0 g/dL Heart Function - Left Ventricular Ejection Fraction (LVEF) ≥ 50% as measured by transthoracic echocardiogram ECHO) All tests must be performed ≤ 3 days prior to study enrollment. Eligibility for hemoglobin count may be reached by transfusion
* Signed and dated informed consent document by the patient, indicating that the patient has been informed of all the pertinent aspects of the trial prior to study enrollment
* Willingness and ability of the patient to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* The patient is active participant in another clinical trial.
* Exclusion of patients in the event of

  * surgery for recurrence/progression within 1 week prior to study enrollment
  * chemotherapy within 4 weeks prior to study enrollment
  * treatment with more than one chemotherapy regime
  * radiation therapy within 8 weeks to study enrollment
  * evidence in baseline MRI of intratumoral or peritumoral hemorrhage deemed clinically significant by the treating physician (area of hemorrhage > 25% of tumor area)
* Significant Co-Morbidities within 12 months prior to study enrollment

  * myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure
  * pulmonary embolus
  * cerebro-vascular accident including TIA (transient ischemic attack)
* Significant Co-Morbidities at Baseline Evaluation

  * Clinically significant ongoing cardiac dysrhythmias of grade ≥ 2, atrial fibrillation of any grade, QTc interval > 470 ms measured by electrocardiogram (ECG)
  * Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
  * A known HIV (human immunodeficiency virus) or Hepatitis B/C infection or severe acute infection
* Anticoagulation: Current treatment with therapeutic doses of Marcoumar / Sintrom excluding thrombosis prophylaxis with low dose Heparin.
* Antiepileptic Drugs: Concurrent use of EIADs within 2 weeks of study enrollment (patients must discontinue EIAD treatment ≥ 14 days prior to study enrollment)
* Pregnancy, Breastfeeding and Non-Contraception

  * Female patients who are pregnant or nursing
  * Patients who are sexually active and unwilling or unable to use a medically acceptable method of contraception during the trial.
* Evidence of increased intracranial pressure

  * midline shift > 5 mm
  * distinct nausea and vomiting
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart excess risk associated with study participation or study drug administration, or which would make the patient inappropriate for entry into this study. The decision to enroll the patient in this study is in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | 6 months after tumor progression
Median time to tumor progression | Time to tumor progression

SECONDARY OUTCOMES:
Overall survival | Time from study inclusion to death
Overall survival rate at 12 months | 12 months after tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Stockhammer, MD, Prof., Principal Investigator — Medical University Innsbruck
Locations (10):
- Austria (6):
  - Paracelsus Medical University, Salzburg, Salzburg
  - LKH Feldkirch, Feldkirch
  - Medical University Innsbruck, Innsbruck
  - LNK Wagner-Jauregg, Linz
  - Kaiser-Franz-Josef Spital Wien, Vienna
  - Medical University Vienna, Vienna
- Germany (4):
  - University Hospital of Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Hospital of Mannheim, Mannheim, Baden-Wurttemberg
  - University Hospital of Bonn, Bonn, North Rhine-Westphalia
  - University Hospital of Berlin, Berlin, State of Berlin

REFERENCES:
- [Derived] Hutterer M, Nowosielski M, Haybaeck J, Embacher S, Stockhammer F, Gotwald T, Holzner B, Capper D, Preusser M, Marosi C, Oberndorfer S, Moik M, Buchroithner J, Seiz M, Tuettenberg J, Herrlinger U, Wick A, Vajkoczy P, Stockhammer G. A single-arm phase II Austrian/German multicenter trial on continuous daily sunitinib in primary glioblastoma at first recurrence (SURGE 01-07). Neuro Oncol. 2014 Jan;16(1):92-102. doi: 10.1093/neuonc/not161. Epub 2013 Dec 4. PMID 24311637
- See also: Homepage of the Medical University Innsbruck — http://www.i-med.ac.at